CLINICAL TRIAL: NCT04138394
Title: VItamin C in Thermal injuRY: The VICToRY Trial A Phase III Multi-center Randomized Trial
Brief Title: VItamin C in Thermal injuRY: The VICToRY Trial
Acronym: VICToRY
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: After the 1st interim analysis, on the recommendation of the DSMC, the steering committee decided to stop enrollment of new patients. The study is ongoing for the currently enrolled patients. More info to follow when available for public disclosure.
Sponsor: Clinical Evaluation Research Unit at Kingston General Hospital (Other)
Collaborators: Dr. Christian Stoppe, MD, Co-Principal Investigator, Wurzburg University, Wurzburg, Germany (Unknown)
Responsible Party: Principal Investigator, Daren K. Heyland, Dr. Daren Heyland, MD, MSc, FRCPC, Clinical Evaluation Research Unit at Kingston General Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VICToRY
Record Dates: First submitted 2019-10-21; First posted 2019-10-24 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Shock; Thermal Burn
MeSH Terms: conditions — Shock | interventions — Ascorbic Acid; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients will be allocated to receive intravenous vitamin C at 50mg/kg, every 6 hrs for 96 hrs or placebo. We justify this proposed dosing strategy as the proposed dose of vitamin C has been shown to be safe and effective in patients with sepsis and lung injury whereas prior dosing strategies used in the burns literature (66 mg/kg/24 hours) have safety issues and are not long enough in duration. Control group: patients will receive a similar amount of placebo (either D5W or saline) delivered in the same manner as the vitamin C.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Allocation will be random and concealed and will be blinded to everyone except the pharmacist at each site. The vitamin C will be sourced locally and prepared in a blinded manner by local research pharmacies that will be responsible for preparing study samples and delivering them to the ICU in a blinded fashion. The randomization system, which has proven reliable in several prior RCTs, has a robust audit trail, and will maintain concealment and blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vitamin C (Experimental): Patients will receive intravenous vitamin C at 50mg/kg every 6 hours for 96 hours
  Interventions: Drug: Ascorbic Acid
- Control group (Placebo Comparator): Patients will receive a similar amount of placebo (either D5W or saline) delivered in the same manner as the vitamin C.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Ascorbic Acid — Patients will receive intravenous vitamin C (50 mg/kg every 6 hours for 96 hours).
  Other Names: vitamin C
  Arms: Vitamin C
Drug: placebo — Patients will receive a similar amount of placebo (either D5W or saline) delivered in the same manner as the vitamin C.
  Other Names: saline; D5W
  Arms: Control group

SUMMARY:
This study aims to show that giving high dose, intravenous vitamin C in addition to standard care to burned critically ill patients will be associated with less organ dysfunction, improved survival and a quicker rate of recovery. In this study, all patients will receive standard care and of the patients will also receive high dose intravenous vitamin C, while the other half of patients will receive placebo.

DETAILED DESCRIPTION:
In certain disease states, such as those associated with severe burns and other critical illnesses, the relationship between nutrient deficiencies, altered immune status, and acquired infection has been recognized for many years. More than in any other injury, the inflammation and catabolism associated with severe burns can exacerbate nutrient deficiencies, thereby predisposing patients to impaired immune function and increased risk of developing infectious complications, organ dysfunction, and death.

We aim to conduct a large-scale, multi-center randomized trial to evaluate the effect of high-dose (50mg/kg every 6 hours for 96 hours) intravenous vitamin C in addition to standard of care (SOC) on 28-days composite outcome of Persistent Organ Dysfunction (POD) and all-cause mortality compared to add-on placebo and SOC.

Patients will be allocated to 2 groups, active or control: patients in the active group will receive intravenous vitamin C at 50mg/kg every 6 hrs for 96 hrs. Patients in the control group will receive a similar amount of placebo (either D5W or saline) delivered in the same manner as the vitamin C. This study will be the first large international multi-centre trial examining the effects of high dose intravenous vitamin C in burn patients. It represents a unique collaboration of burn units worldwide that is coordinated by the Clinical Evaluation Research Unit, based in Kingston Ontario Canada, a coordinating center that has demonstrated the ability to run multi-center trials and translate findings into practice.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Deep 2nd and/or 3rd degree burns requiring skin grafting
* Minimum burn size of ≥ 20% Total Body Surface Area (TBSA)

Exclusion Criteria:

* >24 hours from admission to participating hospital to consent.
* Patients admitted to burn unit >24 from injury or accident.
* Patients who are moribund (not expected to survive the next 72 hours).
* Pregnancy (pregnancy will be ruled out as part of standard of care) or lactating.
* Enrollment in another industry sponsored ICU intervention study.
* Receiving high-dose IV vitamin C already (enteral or oral vitamin C is allowed).
* Known glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* Recent history of kidney stones (within the last year).
* Concomitant use of hydroxycobalamin (vitamin B12) for suspected cyanide poisoning.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 666 (Estimated)
Dates: Start 2020-07-24 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Persistent Organ Dysfunction + Death | at 28 days
  Persistent organ dysfunction (PODS)+death, a novel composite endpoint that combines being alive and being free of organ support (inotropes or vasopressors, renal replacement therapy and mechanical ventilation)
Time to discharge alive from hospital | 90 days
  Time to discharge alive from hospital, a composite of mortality and length of stay is similar to "ventilator- free days", which is a widely accepted and commonly used outcome in intensive care research.

OTHER OUTCOMES:
ICU length of stay | 90 days
  Duration of time in the ICU
Duration of mechanical ventilation | 90 days
  Length of time on mechanical ventilation, including still on mechanical ventilation at time of discharge.
ICU readmission rate | 90 days
  Incidents of readmission to ICU from within the hospital
Hospital mortality | 90 days
  Did the patient die in hospital or was the patient discharged?
Hospital length of stay | 90 days
  Duration of time in the hospital
Wound healing | 90 days
  time-to-95% graft closure
Gram negative bacteremia | 90 days
  Venous or arterial blood cultures that show bacteremia with Gram-negative bacilli
6 month mortality | 6 months
  Is the patient alive or deceased 6 months post admission.
Health-related quality of life | 6 months
  Administration of the SF-36 questionnaire 6 months post admission

CONTACTS AND LOCATIONS:
Overall Officials: Daren K Heyland, MD, Principal Investigator — Queen's University
Locations (33):
- United States (10):
  - Arizona Burn Center Valleywise Health, Phoenix, Arizona
  - Bridgeport Hospital, Bridgeport, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - The University of Chicago Medical Center, Chicago, Illinois
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Mercy Hospital St. Louis, St Louis, Missouri
  - The Ohio State University Medical Center, Ohio City, Ohio
  - University of Texas Health Science Center - Houston, Houston, Texas
  - Harborview Medical Center - Seattle, Seattle, Washington
  - Ascension Columbia St. Mary's, Milwaukee, Wisconsin
- Belgium (4):
  - Grand Hopital de Charleroi, Charleroi, Hainaut
  - Ghent University Hospital, Ghent, Oost Vlaanderen
  - Belgium Military Hospital, Military Hospital, Brussels
  - Centre Hospitalier Universitaire de Liege, Liège
- Canada (5):
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton General Hospital, Hamilton Health Sciences Corporation, Hamilton, Ontario
  - Sunnybrook Health Sciences Centre, Ross Tilley Burn Centre, Toronto, Ontario
  - Centre de recherche du CHUM, Montreal, Quebec
  - CHU de Québec-Université Laval, Hôpital de l'Enfant-Jésus, Québec, Quebec
- Hospital San Juan de Dios, San José, Provincia de San José, Costa Rica
- Germany (6):
  - BG Klinik Tübingen, Tübingen, Baden-Wurttemberg
  - Klinikum St. George, Leipzig, Saxony
  - RWTH Aachen University, Aachen, Aachen
  - Merheim Medical Center, Hospitals of Cologne, Cologne
  - Berufsgenossenschaftliche Unfallklinik Ludwigshafen, Ludwigshafen
  - University Hospital Würzburg, Würzburg
- Hospital Central Dr. Ignacio Morones Prieto, San Luis Potosí City, San Luis Potosí, Mexico
- Centro Nacional del Quemado y Cirugías Reconstructivas, Asunción, Paraguay
- Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand
- United Kingdom (4):
  - Chelsea and Westminster Hospital, Chelsea, London
  - Queen Elizabeth Hospital Birmingham, Birmingham, Mindelsohn Way
  - St Helens and Knowsley Hospitals NHS Trust, Prescot
  - The Mid Yorkshire Hospitals NHS Trust, Wakefield

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT04138394/Prot_SAP_000.pdf